CLINICAL TRIAL: NCT04199221
Title: Use of Stress Inoculation Training in Medical Education
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: lack of enrollment
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HM20014865
Record Dates: First submitted 2019-12-11; First posted 2019-12-13 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2023-12

CONDITIONS: Stress
Keywords: Stress Inoculation; Medical Education; Simulation Training

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Lecture (No Intervention): an initial brief lecture with no further training
- Stress management (Experimental): an initial brief lecture with stress management lecture
  Interventions: Behavioral: Stress Innoculation Training (SIT)
- Hands-on training (Active Comparator): an initial brief lecture with addition hands-on training for the task
  Interventions: Behavioral: Extra attempt
- Stress management and hands-on training (Experimental): an initial brief lecture with both stress management lecture and additional hands-on training
  Interventions: Behavioral: Stress Innoculation Training (SIT); Behavioral: Extra attempt

INTERVENTIONS:
Behavioral: Stress Innoculation Training (SIT) — 1 hour lecture that will cover the conceptualization phase and skills-training phase portions of stress inoculation training.
  Arms: Stress management; Stress management and hands-on training
Behavioral: Extra attempt — an extra attempt at intubating a mannequin configured at a difficulty level higher than will be used in the future scenarios
  Arms: Hands-on training; Stress management and hands-on training

SUMMARY:
The purpose of this research study is to test the feasibility and effectiveness of SIT in teaching medical students to perform in high-fidelity simulation settings similar to those they may experience in their practice.

DETAILED DESCRIPTION:
This is a study examining stress inoculation training and its potential role in medical education. The medical field exposes students and providers to various stressful situations each and every day. Various organizations including military organizations have introduced concepts of stress inoculation training (SIT) to help learners manage these situations to produce optimal performance.

ELIGIBILITY:
Inclusion Criteria:

* 1st and 2nd year medical students who are at least 18 years old

Exclusion Criteria:

* Prior airway management experience (including but not limited to former medics, respiratory technicians, CRNAs)
* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2021-08-26 (Actual); Primary Completion 2023-12-29 (Actual); Study Completion 2023-12-29 (Actual)

PRIMARY OUTCOMES:
Change in anxiety - visual analog | Baseline to up to 3 weeks
  Change in anxiety will be assessed using the Visual Anxiety Scale (VAS/VAS-A), a widely used scale that has been validated in multiple settings to detect changes in anxiety level. A 10cm line will be drawn on the screen and participants will be asked to rate their level of anxiety by clicking somewhere on the line - the leftmost portion coinciding with no anxiety, the rightmost portion coinciding with extreme anxiety. Each millimeter to the right of the initial start of the line counts as 1 point out of 100.
Change in state-trait anxiety | Baseline to up to 3 weeks
  Spielberger State-Trait Anxiety Inventory 6 (STAI-6) will be used to measure state-trait anxiety. The STAI-6 is a validated 6-question form of the STAI-Y, a commonly used and validated measure of anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Nathan J Lewis, MD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No